CLINICAL TRIAL: NCT04373135
Title: A Study to Evaluate Health Behavior and Access Impacts Due to COVID-19 and for Community Engagement of Stakeholders Surrounding Scarce Resource Allocation Policy.
Brief Title: Understanding Community Considerations, Opinions, Values, Impacts, and Decisions for COVID-19
Acronym: UC-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Russell G. Buhr, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLA-20-000683
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-05

CONDITIONS: Covid-19; Critical Illness; Attitude of Health Personnel; Attitude to Health; Health Behavior; Health Care Utilization
Keywords: health disparity; scarce resource allocation; triage; community engagement
MeSH Terms: conditions — COVID-19; Critical Illness; Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Pre-/post-intervention survey with random allocation of a brief educational intervention about scarce resource allocation policy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Subjects will be provided a brief educational intervention prior to completing follow up survey about SRA attitudes and knowledge
  Interventions: Behavioral: Brief educational video
- Control (No Intervention): Subjects will not be provided any prior to completing follow up survey about SRA attitudes and knowledge

INTERVENTIONS:
Behavioral: Brief educational video — A brief educational video will be displayed explaining the mechanics of how SRA policies operate, how they are decided, and what patients' and healthcare workers' rights are surrounding them.
  Arms: Experimental

SUMMARY:
The novel coronavirus (COVID-19) is affecting the way many people live their lives, including seeking medical care and maintaining good self-care to keep healthy. Additionally, in the event many people become critically ill at once, COVID-19 has the possibility of overwhelming hospitals to the point where they have to make decisions about how to determine who receives intensive care and life-support measures. Many hospitals as well as local or state governments have been working on policies to determine how to make these decisions. This study seeks to learn about how COVID-19 has affected the way patients and healthcare providers care for themselves and about their thoughts and concerns about policies that may "ration" life-support resources.

DETAILED DESCRIPTION:
Background:

COVID-19 has led to significant disruptions to usual operations of the health care system and routines of millions of people. Regular medical appointments have been preempted or converted to telemedicine, dietary changes have occurred due to food supply chain strain, and exercise regimens altered by physical distancing policies, all of which may affect preventive care and chronic illness management. Additionally, anxiety about risk of developing COVID-19 and the availability of health care resources may alter care-seeking behaviors even for serious conditions, e.g., heart attacks.

Understanding personal health and protective behaviors under threat of COVID-19 is an epidemiologic imperative and can inform immediate public health response as well as planning for population health needs post-crisis.

Critical care capacity during COVID-19 is also a matter of extreme concern. Limitations in capacity, particularly mechanical ventilators have necessitated scarce resource allocation (SRA) policies, which outline triage protocols while observing ethical principles of distributive justice, transparency, and equitability.

In practice, these policies determine which patients are most likely to benefit from intensive care, and some patients with a significantly heightened risk for mortality are less likely to be prioritized in critical care allocation decisions. The uncertainty around prioritization and threat of rationing of care has generated public attention and anxiety evident in medical journals, news outlets, and on social media.

The rapidity of this crisis has compelled rapid development and/or modification of SRA policies without the rigorous stakeholder engagement or evaluations of acceptance of these policies by both laypersons and practitioners tasked with implementing such policies. Two states (CA & NY), among the most affected by COVID-19, have recently developed new SRA policies, creating a unique opportunity to evaluate how these policies are understood and perceived by the patients most likely to be impacted by them and the practitioners who will implement them. Moreover, given the complexity of the ethical underpinnings and potential misinformation about SRA policies, there is a clear need to determine if a brief educational intervention can influence perception and knowledge about these containment and management policies.

The investigators propose to undertake rapid recruitment of a national cohort of individuals and health care workers to understand knowledge and perceptions of public health and clinical efforts during this evolving pandemic; and to implement a randomized controlled trial within this cohort to test the ability of a brief intervention to improve knowledge and perceptions about the health care system's capacity to provide equitable care during a pandemic. The specific aims are to:

* Aim 1: Determine how key indicators of population health (including health status, health behaviors, and access to care) have changed during the COVID-19 outbreak in the US.
* Aim 1a: Uncover the extent of racial/ethnic and socioeconomic disparities in the impacts of COVID-19 on health, health behaviors, and access to care.
* Aim 2: Assess the public's and practitioners' knowledge and values around SRA policies and examine which individual characteristics correlate with these knowledge and values.
* Aim 3: Evaluate the impact of a brief educational intervention on knowledge and values for SRA policy among the public and health care workers.

Population & Recruitment:

For Aim 1, the investigators will employ national outreach strategies via social media and partnerships with national organizations to recruit a sample of adults (ages 18 and older) from the general population. The investigators will enrich this sample by direct recruitment efforts (via online health portal invitation) of over 300,000 patients in the Southern California Area who are cared for in the University of California at Los Angeles Health System (UCLA Health).

For Aim 2, the investigators will employ similar national outreach strategies involving professional language targeted posts on social media sites (e.g., Doximity, LinkedIn) to recruit a sample of health care providers. Additionally, this cohort will be enriched by direct recruitment efforts of health workers employed by UCLA. Cohort participants in Aims 1 & 2 from California and New York (residence determined based on ZIP code) will be randomized for Aim 3 to receive either a brief educational video or no intervention. All participants (Aims 1-3) will be invited to complete three surveys (baseline, one-month post-intervention follow-up, and four-month follow-up; Figure 1). Sample recruitment path and representativeness with be assessed using unique source links and standard visitor tracking analytics built into the study website.

Survey Assessments: Participants will first be presented with an online consent form that includes language typical of a written consent and upon affirming consent will be directed to complete the baseline survey. The patient baseline survey will collect sociodemographic information (including ZIP code), chronic conditions and current health status, health behaviors, anxiety and stress levels, changes to health and care seeking behaviors (e.g., social distancing, medication adherence, care-seeking behaviors), and will include series of questions assessing perceptions and attitudes and knowledge about SRA policies and how they are implemented (e.g., values about how decisions are made, understanding of prioritization versus exclusion from critical care). Demographic, behavioral, and access questions are largely derived from the validated Behavioral Risk Factor Surveillance System questionnaires which will provide a historical comparison for study results. For providers, additional questions about the characteristics of the provider will include specialty, years of practice, and trainee status. Follow-up surveys will re-administer key baseline questions on SRA knowledge and values, personal health behaviors, and COVID-19-specific impacts (e.g., if they or a loved one was hospitalized and/or was subject to an SRA policy decision, and for providers, whether they had to use an SRA tool during their practice); follow-up surveys will additional ascertain exposure to media coverage about COVID-19 and SRAs in the intervening windows. All surveys will be administered via Research Electronic Data Capture (REDCap) system and links to complete follow-up surveys will be automatically delivered to participants via e-mail, with up to four reminders to complete, facilitating linkage between survey administration within individuals. E-mails will be stored separately from survey data in REDCap and will be permanently deleted upon study completion.

Intervention and Randomization: The investigators will develop a brief (~3 min) video intervention that describes what SRA policies are, how they were developed, who is most likely to be impacted, and patients' rights under these policies. Two versions will be utilized, one oriented for a lay audience and one for practitioners using technical medical language, but both will be relevant to the policies currently in place in two of the hardest hit states (NY and CA). The investigators have contracted with WorldWise Productions, who have completed similar videos for multiple other UCLA Health and DGSOM projects. The intervention will be hosted on a private YouTube channel and embedded in REDCap so that it can be automatically delivered as part of the survey. The investigators will execute a stratified randomization scheme based on state, age, and education level to allocate respondents from CA and NY evenly between intervention and control. Participants outside CA & NY will serve as negative controls. All participants will receive a post-intervention survey with repeat assessment (as described above).

Focus Groups:

Because COVID-19 is a rapidly evolving crisis and there are no pre-existing validated questions to ascertain COVID-19 perceptions and impacts, the investigators plan to conduct a final qualitative follow-up (post-crisis) with a geographically and sociodemographically diverse selection of participants (both patients and providers) in order to obtain a more nuanced and complete examination of perceptions, attitudes, and experiences. Participants selected will be invited to participate approximately 4-6 months later (after the COVID-19 crisis has slowed). Key health behavior themes will include experience with telemedicine, disruptions to health care access, and general changes to health during and after COVID-19 pandemic; particular attention will be paid to inequities in these outcomes. Key SRA themes will include the method of selecting patients, concerns about equity, special considerations for disadvantaged or vulnerable populations, and perceptions of the crisis response in general. Groups will be conducted via web-conference using Zoom and recorded, transcribed, and then qualitative methods used to analyze transcripts for key themes. The investigators plan to conduct approximately 15 focus groups of 5-10 participants each.

Power:

To detect a ½ standard deviation change in the number of correct knowledge items between the intervention and control arms with 90% power and a two-sided α=0.05, 172 total participants are needed to complete follow-up. Based on prior work with >80% trial retention and recruitment of 55 participants per day, the investigators anticipate recruiting the necessary 216 baseline trial participants within 4 days. The investigators anticipate that they will substantially exceed the targets to achieve desired trial power.

Milestones & Actionable Outcomes:

There is a paucity of evidence on changes in health status and behaviors related to physical distancing policies and the widescale adoption and implementation of SRA policies. By determining how health behaviors and access to care are impacted at baseline, the investigators can directly issue recommendations for patients and providers aimed at affecting population health and mitigating disparities therein. The assessment of SRA policies and how they are perceived and implemented during a crisis will dramatically increase the ability to design and apply such policies in a fair and equitable way and to determine what adjustments to the policies from a clinical perspective are needed to ensure that disproportionate burden is not borne by vulnerable patients. As the baseline survey has already been developed, piloted, and programmed into REDCap and the investigators have established partnerships with several organizations who have already agreed to assist with study recruitment - the investigators are prepared to initiate the study immediately. Production on the intervention video can begin as soon as notice of funds have been received. Trial milestones include recruitment of >216 participants from CA & NY within the first week of recruitment and retention of >172 participants at one-month follow-up. Additional milestones include the submission of several research papers to high-impact medical journals detailing research findings.

ELIGIBILITY:
Inclusion Criteria:

* Participants shall be adults aged 18 years or older
* Willingness and ability to participate in an internet-based survey

Exclusion Criteria:

* Children under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1971 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement in knowledge surrounding SRA policy | 1 month, 6 months
  Improvement in knowledge item score of 1/2 SD points on follow up after intervention delivery and at final follow up
Stability of in anxiety surrounding SRA policy | 1 month, 6 months
  No worsening in anxiety scale of 1/2 SD responses on follow up after intervention delivery and at final follow up
Improvement in trust surrounding SRA policy | 1 month, 6 months
  Improvement in trust scale of 1/2 SD on follow up after intervention delivery and at final follow up

CONTACTS AND LOCATIONS:
Overall Officials: Russell G Buhr, MD, PhD, Principal Investigator — Division of Pulmonary & Critical Care Medicine, UCLA; Lauren E Wisk, PhD, Principal Investigator — Division of General Internal Medicine & Health Services Research, UCLA
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data requests for analysis may be approved by the investigators upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 4 months of study closure
Access Criteria: Reasonable request to investigators

REFERENCES:
- [Background] Rundle AG, Park Y, Herbstman JB, Kinsey EW, Wang YC. COVID-19-Related School Closings and Risk of Weight Gain Among Children. Obesity (Silver Spring). 2020 Jun;28(6):1008-1009. doi: 10.1002/oby.22813. Epub 2020 Apr 18. No abstract available. PMID 32227671
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Powell T, Christ KC, Birkhead GS. Allocation of ventilators in a public health disaster. Disaster Med Public Health Prep. 2008 Mar;2(1):20-6. doi: 10.1097/DMP.0b013e3181620794. PMID 18388654
- [Background] Truog RD, Mitchell C, Daley GQ. The Toughest Triage - Allocating Ventilators in a Pandemic. N Engl J Med. 2020 May 21;382(21):1973-1975. doi: 10.1056/NEJMp2005689. Epub 2020 Mar 23. No abstract available. PMID 32202721
- [Background] Emanuel EJ, Persad G, Upshur R, Thome B, Parker M, Glickman A, Zhang C, Boyle C, Smith M, Phillips JP. Fair Allocation of Scarce Medical Resources in the Time of Covid-19. N Engl J Med. 2020 May 21;382(21):2049-2055. doi: 10.1056/NEJMsb2005114. Epub 2020 Mar 23. No abstract available. PMID 32202722
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Yang J, Zheng Y, Gou X, Pu K, Chen Z, Guo Q, Ji R, Wang H, Wang Y, Zhou Y. Prevalence of comorbidities and its effects in patients infected with SARS-CoV-2: a systematic review and meta-analysis. Int J Infect Dis. 2020 May;94:91-95. doi: 10.1016/j.ijid.2020.03.017. Epub 2020 Mar 12. PMID 32173574
- [Background] Antommaria AHM, Gibb TS, McGuire AL, Wolpe PR, Wynia MK, Applewhite MK, Caplan A, Diekema DS, Hester DM, Lehmann LS, McLeod-Sordjan R, Schiff T, Tabor HK, Wieten SE, Eberl JT; Task Force of the Association of Bioethics Program Directors. Ventilator Triage Policies During the COVID-19 Pandemic at U.S. Hospitals Associated With Members of the Association of Bioethics Program Directors. Ann Intern Med. 2020 Aug 4;173(3):188-194. doi: 10.7326/M20-1738. Epub 2020 Apr 24. PMID 32330224
- [Background] Daugherty Biddison EL, Faden R, Gwon HS, Mareiniss DP, Regenberg AC, Schoch-Spana M, Schwartz J, Toner ES. Too Many Patients...A Framework to Guide Statewide Allocation of Scarce Mechanical Ventilation During Disasters. Chest. 2019 Apr;155(4):848-854. doi: 10.1016/j.chest.2018.09.025. Epub 2018 Oct 11. PMID 30316913
- [Background] Biddison ELD, Gwon HS, Schoch-Spana M, Regenberg AC, Juliano C, Faden RR, Toner ES. Scarce Resource Allocation During Disasters: A Mixed-Method Community Engagement Study. Chest. 2018 Jan;153(1):187-195. doi: 10.1016/j.chest.2017.08.001. Epub 2017 Aug 9. PMID 28802695
- [Background] Biddison LD, Berkowitz KA, Courtney B, De Jong CM, Devereaux AV, Kissoon N, Roxland BE, Sprung CL, Dichter JR, Christian MD, Powell T; Task Force for Mass Critical Care; Task Force for Mass Critical Care. Ethical considerations: care of the critically ill and injured during pandemics and disasters: CHEST consensus statement. Chest. 2014 Oct;146(4 Suppl):e145S-55S. doi: 10.1378/chest.14-0742. PMID 25144262
- [Background] Wisk LE, Nelson EB, Magane KM, Weitzman ER. Clinical Trial Recruitment and Retention of College Students with Type 1 Diabetes via Social Media: An Implementation Case Study. J Diabetes Sci Technol. 2019 May;13(3):445-456. doi: 10.1177/1932296819839503. Epub 2019 Apr 22. PMID 31010315
- [Background] Pierannunzi C, Hu SS, Balluz L. A systematic review of publications assessing reliability and validity of the Behavioral Risk Factor Surveillance System (BRFSS), 2004-2011. BMC Med Res Methodol. 2013 Mar 24;13:49. doi: 10.1186/1471-2288-13-49. PMID 23522349
- [Derived] Buhr RG, Huang CX, Romero R, Wisk LE. Bolstering agreement with scarce resource allocation policy using education: a post hoc analysis of a randomized controlled trial. BMC Health Serv Res. 2025 Apr 14;25(1):540. doi: 10.1186/s12913-025-12712-x. PMID 40229711
- [Derived] Buhr RG, Romero R, Wisk LE. Promotion of Knowledge and Trust Surrounding Scarce Resource Allocation Policies: A Randomized Clinical Trial. JAMA Health Forum. 2024 Oct 4;5(10):e243509. doi: 10.1001/jamahealthforum.2024.3509. PMID 39422889
- [Derived] Loui HF, Li J, Jackson NJ, Romero R, Wisk LE, Buhr RG. Tobacco consumption behavior change during the COVID-19 pandemic is associated with perceived COVID threat. BMC Public Health. 2024 Oct 15;24(1):2827. doi: 10.1186/s12889-024-20259-5. PMID 39407204
- [Derived] Wisk LE, Buhr RG. Rapid deployment of a community engagement study and educational trial via social media: implementation of the UC-COVID study. Trials. 2021 Aug 2;22(1):513. doi: 10.1186/s13063-021-05467-3. PMID 34340693
- [Derived] Wisk LE, Buhr RG. Rapid Deployment of A Community Engagement Study And Educational Trial Via Social Media: Implementation of The UC-COVID Study. Res Sq [Preprint]. 2021 May 7:rs.3.rs-359099. doi: 10.21203/rs.3.rs-359099/v1. PMID 34013254